CLINICAL TRIAL: NCT06925100
Title: A Multicenter, Prospective, Phase IV, Interventional Study to Investigate the Effectiveness and Safety of Bempedoic Acid in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia in Taiwan - The CLEAR Taiwan Study
Brief Title: A Study to Investigate the Effectiveness and Safety of Bempedoic Acid in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia in Taiwan
Acronym: CLEAR Taiwan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA-TWMA-HLD-4001
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Primary Hypercholesterolemia or Mixed Hyperlipidemia
Keywords: Taiwan; low-density lipoprotein cholesterol; primary hypercholesterolemia; bempedoic acid; mixed dyslipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bempedoic acid (Experimental): 180 mg, oral, once daily for 12 weeks
  Interventions: Drug: Bempedoic acid 180 mg tablet

INTERVENTIONS:
Drug: Bempedoic acid 180 mg tablet — 180 mg tablet, once daily administered for 12 weeks

SUMMARY:
Cardiovascular disease (CVD) is a chronic non-communicable disease among the most common causes of death worldwide. Substantial reductions in risks of CVD can be achieved through the management of modifiable risk factors, particularly low-density lipoprotein cholesterol (LDL-C). However, only 18.3% of high-risk primary prevention patients and 20.7% of secondary prevention patients achieved the treatment goals based on the 2019 ESC guidelines. Similar trends were reported by the latest European multinational observational SANTORINI study. These real-world evidence data indicate the suboptimal implementation of ESC/EAS 2019 guidelines on LDL-C, particularly the low use of combinational lipid-lowering therapy (LLT), leading to a substantial proportion of patients remaining at high residual risk of ASCVD events.

Bempedoic acid, a first-in-class novel nonstatin lipid-lowering agent, was approved by the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA) in 2020 for the treatment of primary hypercholesterolemia. Bempedoic acid inhibits cholesterol biosynthesis through the inhibition of adenosine triphosphate-citrate lyase, an upstream enzyme of 3-hydroxy-3-methylglutaryl-coenzyme A reductase. The unique hepatic activation of bempedoic acid results in limited exposure to skeletal muscle, which prevents musculoskeletal-related adverse events.

Phase II and III RCTs have demonstrated efficacy with adequate safety data of bempedoic acid as mono- or combination therapy with statins and ezetimibe. The CLEAR outcomes trial demonstrated the benefit of bempedoic acid in lowering the risks of major adverse cardiovascular events in statin-intolerant patients.

However, there is limited data on bempedoic acid treatment in East Asian subjects and no data in the Taiwanese population, despite modeling data from large studies indicating the potential for no ethnic differences. To investigate the effectiveness and safety of bempedoic acid in a Taiwanese population, this phase IV study is conducted to examine the treatment outcomes in approximately 180 patients using bempedoic acid in Taiwan.

DETAILED DESCRIPTION:
This is a multicenter, prospective, phase IV, single-arm, interventional study investigating the effectiveness and safety of bempeodoic acid in Taiwanese patients with hypercholesterolemia or mixed dyslipidemia. The study will be conducted in three medical centers in Taiwan to include approximately 180 patients with hypercholesterolemia or mixed dyslipidemia.

All enrolled patients will receive bempedoic acid 180 mg once daily for 12 weeks, with a total of 3 visits as follows: Baseline, Week 4, and Week 12; and there will be one follow-up visit at 2 to 4 weeks after discontinuation for those who discontinue the study due to adverse events. Across the study period, all patients must maintain the regimen (including medication, dose, and frequency) of their background LLT that they received before initiating bempedoic acid treatment.

Aside from bempedoic acid, LLT, study visits, and assessments, other medical procedures and prescriptions will be based on physicians' judgments per real-world clinical practice. Subjects will be continually followed up from the enrollment date until Week 12, bempedoic acid discontinuation, study discontinuation, or lost to follow-up, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Diagnosed with primary hypercholesterolemia (heterozygous familial and non-familial) or mixed dyslipidemia:

   * Patients who have been on statin or statin combining with other lipid-lowering therapies* (both under the maximum tolerated dose of statin) for at least 4 weeks, but unable to reach LDL-C goals† OR
   * Patients who are statin-intolerant or contraindicated to statin, alone or have been on other non-statin lipid-lowering therapies* for at least 4 weeks, but unable to reach LDL-C goals†

     * Other lipid-lowering therapies: Ezetimibe, Cholesterol and/or bile acid, absorption inhibitors, PCSK9 inhibitors, Omega-3 fatty acids, Fibrates, or Niacin derivatives

     † LDL-C goals are defined as:
   * Patients with ASCVD or had conducted coronary revascularization procedures (e.g., PCI or CABG): LDL-C < 70 mg/dL
   * Patients aside from the above population: LDL-C < 100 mg/dL
3. The physician intends to prescribe bempedoic acid per locally approved label (the study intends no intervention in physicians' judgement on the prescription of bempedoic acid)
4. Provide written informed consent

Exclusion Criteria:

1. Concurrent participation in an interventional study (simultaneous participation in other non-interventional studies is acceptable)
2. With eGFR < 30 mL/min/1.73 m2, end-stage renal disease (ESRD) on dialysis, severe hepatic impairment (Child-Pugh C), bempedoic acid contraindications (i.e., hypersensitivity to the active substance or any of the excipients, galactose intolerance, pregnancy, breastfeeding, concomitant use with simvastatin > 40 mg daily)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in LDL-C level at Week 12 | 12 weeks
  To investigate the percentage change from baseline in LDL-C level at Week 12

SECONDARY OUTCOMES:
LDL-C goal attainment rate at Week 12 | 12 weeks
  To investigate the LDL-C goal attainment rate at Week 12, the LDL-C goal is set as follows:
  1. Patients with ASCVD or had conducted coronary revascularization procedures (e.g., PCI or CABG): Attainment rate at LDL-C < 100 mg/dL, LDL-C < 70 mg/dL, and LDL-C < 55 mg/dL
  2. Patients aside from the above population: Attainment rate at LDL-C < 100 mg/dL
Percentage change from baseline in other lipid parameters (total cholesterol [TC], apolipoprotein B [apoB], high-density lipoprotein cholesterol [HDL-C], non-HDL-C, and triglycerides [TGs]) at Week 12 | 12 weeks
  To investigate the percentage change from baseline in other lipid parameters (TC, apoB, HDL-C, non-HDL-C, and TG) at Week 12
Percentage change from baseline in hsCRP level at Week 12 | 12 weeks
  To investigate the percentage change from baseline in hsCRP level at Week 12
Adverse events, adverse events of special interest (AESI), and adverse drug reactions associated with bempedoic acid | 12 weeks
  To assess the adverse events, adverse events of special interest (AESI), and adverse drug reactions associated with bempedoic acid

OTHER OUTCOMES:
Percentage change from baseline in lipoprotein A [Lp(a)] at Week 12 | 12 weeks
  To investigate the percentage change from baseline in Lp(a) at Week 12
Change from baseline in HbA1c level at Week 12 | 12 weeks
  To investigate the absolute change from baseline in HbA1c level at Week 12

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/